CLINICAL TRIAL: NCT00800280
Title: A Phase 1, Open-Label, Randomized, Cross-Over Study To Estimate The Effects Of Steady-State Cimetidine On The Pharmacokinetics Of A Single Dose Of PD 0332334 In Healthy Subjects
Brief Title: Evaluating The Effects Of Cimetidine On The Elimination Of PD 0332334 From The Body
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A5361030
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: cimetidine, PD 0332334, organic cation transporter, OCT2, pharmacokinetics
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin; Cimetidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose PD 0332334 (Experimental)
  Interventions: Drug: PD 0332334
- Single dose PD 0332334 with steady-state cimetidine (Experimental)
  Interventions: Drug: PD 0332334; Drug: cimetidine

INTERVENTIONS:
Drug: PD 0332334 — Single 300 mg dose of PD 0332334 immediate release capsules administered orally
  Other Names: imagabalin
  Arms: Single dose PD 0332334
Drug: PD 0332334 — Single 300 mg dose of PD 0332334 immediate release capsules administered orally on Day 2.
  Arms: Single dose PD 0332334 with steady-state cimetidine
Drug: cimetidine — 600 mg q 6 hours cimetidine immediate release formulation administered orally on Days 1 through 5.
  Arms: Single dose PD 0332334 with steady-state cimetidine

SUMMARY:
The purpose of this study is to estimate the effects of multiple doses of cimetidine on the pharmacokinetics of a single dose of PD 0332334 and to evaluate the safety and tolerability of PD 0332334 when co-administered with cimetidine.

DETAILED DESCRIPTION:
Detailed Description:

Additional Study Purpose Details: Evaluate the effects of multiple doses of cimetidine on the pharmacokinetics (e.g., elimination from the body) of a single dose of PD 0332334.

On February 18th 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* male or female adults

Exclusion Criteria:

* Current or history of clinically significant medical illness
* Smokers
* Illicit drug use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
PD 0332334 area under the curve (AUC) from 0 to infinity (AUCinf) | 4 to 6 days
PD 0332334 AUC from 0 to last quantifiable concentration (AUClast) | 4 to 6 days
Half-life (t1/2) of PD 0332334 | 4 to 6 days
Maximum plasma concentration (Cmax) of PD 0332334 | 4 to 6 days

SECONDARY OUTCOMES:
Evaluate the incidence, duration and severity of adverse events | 4 to 6 days
Evaluate the discontinuation due to adverse events | 4 to 6 days
Clinical safety labs | 4 to 6 days
ECG | 4 to 6 days
Vital signs | 4 to 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361030&StudyName=Evaluating%20The%20Effects%20Of%20Cimetidine%20On%20The%20Elimination%20Of%20PD%200332334%20From%20The%20Body